CLINICAL TRIAL: NCT05560035
Title: Effects of Intravenous Lidocaine on Serum THBS2, MMPS and VEGF-C in Patients Undergoing Radical Hyterectomy Surgery After General Anesthesia
Brief Title: The Effect of Intravenous Lidocaine on THBS2 and Angiogenic Factors Expression in Women Undergoing Cervical Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: maling20220922
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Cervical Cancer; Metastatic Cancer
Keywords: Cervical cancer; Tumor progression; Lidocaine; Metalloproteinases; vascular endothelial growth factor; epidermal growth factor; thrombospondin2
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasm Metastasis; Disease Progression | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): Intravenous bolus of 1.5 mg/kg of lidocaine followed by a continuous infusion of 3.0 mg/kg for the first hour, 1.5 mg/kg for the second hour, 0.7 mg/kg for the next 22h.
  Interventions: Drug: Lidocaine
- Normal saline (Placebo Comparator): Normal saline administered as a bolus and an infusion with identical volume and rate changes as the treatment group.
  Interventions: Other: Normal saline (NS)

INTERVENTIONS:
Drug: Lidocaine — Intravenous bolus of 1.5 mg/kg of lidocaine followed by a continuous infusion of 3.0 mg/kg for the frst hour, 1.5 mg/kg for the second hour, 0.7 mg/kg for the next 22h.
  Arms: Lidocaine
Other: Normal saline (NS) — Patients are received equal volumes of saline intravenously until the end of the surgery
  Arms: Normal saline

SUMMARY:
The purpose of this study is to investigate the efficacy of intravenous lidocaine on THBS2, MMPs and VEGF-C in serum in cervical cancer patients undergoing radical hysterectomy under general anesthesia.

DETAILED DESCRIPTION:
The surgical stress response to tumour removal causes bloodstream release of a variety of pro-inflammatory cytokines and other molecules which may affect perioperative immune response and other conditions conducive to residual tumour cell survival that could later emerge as clinical recurrences or metastasis. Lidocaine has analgesic and anti-inflammatory effects, and may also have specific anticancer properties.

Blood serum expression of these molecules (metalloproteinases, vascular endothelial growth factor [VEGF], epidermal growth factor）, play a important role in the metastatic process and tumor progression. lidocaine could affect the course and growth of metastatic tumors by changing the cancer cells, the tumor microenvironment, or both.

We tested the hypothesis that women undergoing cervical cancer resection with these techniques (intravenous lidocaine) have reduced postoperative serum expression of metastasis biomarkers, and may change the outcomes of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients were scheduled by following cervical cancer surgery under general anesthesia
* Aged 18-65 years
* ASA physical status Ⅱ-Ⅲ

Exclusion Criteria:

* Severe heart, pulmonary, hepatic and renal insufficiency
* History of neurological diseases
* Autoimmune disorders
* Antiarrhythmic drugs (amiodarone, verapamil, propafenone)
* Patients' decision to withdraw anytime from the study, and refusal to participate before surgery and at postoperative follow-up
* Allergy to one of the used medications
* Psychiatric illness, psychological disorder, and drug or alcohol abuse
* Unwillingness to comply with the protocol or procedures
* Preoperative treatment of chemotherapy, radiation, NSAID and hormonal therapy
* History of anesthesia and surgery in two weeks
* Coexisting other cancers and intraoperative presence of liver metastasis
* Perioperative treatment of blood transfusion

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline THBS2 before anaesthetic induction and 48 hours after surgery | Baseline and 48 hours after operation
  Blood samples (5 ml) were drawn from each patient before anaesthetic induction, at the end of the operation, 24h and 48 h after operation
Changes from Baseline MMP-2 before anaesthetic induction and 48 hours after surgery | Baseline and 48 hours after operation
  Blood samples (5 ml) were drawn from each patient before anaesthetic induction, at the end of the operation, 24h and 48 h after operation
Changes from Baseline MMP-9 before anaesthetic induction and 48 hours after surgery | Baseline and 48 hours after operation
  Blood samples (5 ml) were drawn from each patient before anaesthetic induction, at the end of the operation, 24h and 48 h after operation
Changes from Baseline VEGF-C before anaesthetic induction and 48 hours after surgery | Baseline and 48 hours after operation
  Blood samples (5 ml) were drawn from each patient before anaesthetic induction, at the end of the operation, 24h and 48 h after operation

SECONDARY OUTCOMES:
Monitoring the severity of postoperative pain with verbalre sponse pain score during the first 48hours postoperatively | at the end of operation and 48 hours after operation
  the severity of pain measured using Visual Analogue Score (VAS) on postoperative days at the moment, 12, 24 and 48 hours after surgery
Resumption of bowel function | at the end of operation and 48 hours after operation
  Record the time to first flatus and the first defecation

OTHER OUTCOMES:
Demographic and anesthetic data, as well as surgical data from each enrolled patient, will be registered on a data collection sheet. | Baseline and 48 hours after operation
  Record the patients demographic and the data of anesthetic and surgical, analysis the connection with primary outcomes